CLINICAL TRIAL: NCT01451164
Title: A Dose-finding Trial of OPC-34712 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-10-002; JapicCTI-111631 (Other: JAPIC)
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2016-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High dose (Experimental)
  Interventions: Drug: OPC-34712
- Mid dose (Experimental)
  Interventions: Drug: OPC-34712
- Low dose (Experimental)
  Interventions: Drug: OPC-34712
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-34712 — orally administered once daily
  Arms: High dose
Drug: OPC-34712 — orally administered once daily
  Arms: Mid dose
Drug: OPC-34712 — orally administered once daily
  Arms: Low dose
Drug: Placebo — orally administered once daily
  Arms: Placebo

SUMMARY:
To investigate the efficacy and safety of OPC-34712 in comparison with placebo in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older to less than 65 years (at time of informed consent) diagnosed with schizophrenia based on DSM-IV-TR diagnostic criteria
* Patients who are hospitalized, or judged to required hospitalization, for acute relapse of schizophrenia at time of informed consent
* Patients who are experiencing acute exacerbation of psychotic symptoms

Exclusion Criteria:

* Female patients who are breastfeeding or who have a positive pregnancy test (urine) result prior to receiving investigational medicinal product
* Patients presenting a first episode of schizophrenia based on the clinical judgment of the investigator
* Patients who are diagnosed with a disease other than schizophrenia (schizoaffective disorder, major depressive disorder, bipolar disorder, posttraumatic stress disorder, anxiety disorder, delirium, dementia, amnesia, or other cognitive disorder) based on current DSM-IV-TR Axis Ι criteria, or who are diagnosed with a personality disorder (borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: kyoji Imaoka, Operating Officer, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kanto Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Brexpiprazole 1mg: Brexpiprazole 1 mg tablet once daily for 6 weeks.
- Brexpiprazole 2mg: Brexpiprazole 2 mg tablet once daily for 6 weeks.
- Brexpiprazole 4mg: Brexpiprazole 4 mg tablet once daily for 6 weeks.
- Placebo: Placebo tablet once daily for 6 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Started | 115 | 115 | 113 | 116
Completed | 72 | 81 | 68 | 70
Not Completed | 43 | 34 | 45 | 46
Not completed — Adverse Event | 19 | 12 | 18 | 21
Not completed — Withdrawal Criteria | 1 | 1 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 14 | 11 | 16 | 17
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 7 | 9 | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo | Total
Number analyzed (Participants) | 115 | 115 | 113 | 116 | 459
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 115 | 115 | 113 | 116 | 459
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (11.5) | 43.3 (12.0) | 44.1 (11.9) | 45.0 (11.9) | 44.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 54 | 58 | 65 | 241
  Male | 51 | 61 | 55 | 51 | 218
Region of Enrollment [Number; unit: participants]
  Japan | 115 | 115 | 113 | 116 | 459

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: Efficacy sample（FAS : Full Analysis Set） consisted of all participants who received at least one dose of study medication and have Baseline and at least one Post-Baseline PANSS total score evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Number analyzed (Participants) | 112 | 113 | 109 | 113
units on a scale
  Week1: number analyzed (Participants) | 110 | 112 | 109 | 113
  Week1 | -2.68 (1.04) | -4.59 (1.03) | -3.42 (1.05) | -3.09 (1.03)
  Week2: number analyzed (Participants) | 94 | 104 | 97 | 98
  Week2 | -5.07 (1.36) | -7.93 (1.33) | -6.80 (1.36) | -4.54 (1.34)
  Week3: number analyzed (Participants) | 86 | 97 | 88 | 85
  Week3 | -6.92 (1.60) | -11.00 (1.55) | -9.42 (1.59) | -6.00 (1.58)
  Week4: number analyzed (Participants) | 80 | 92 | 82 | 77
  Week4 | -8.40 (1.81) | -12.35 (1.74) | -11.21 (1.80) | -5.67 (1.80)
  Week5: number analyzed (Participants) | 76 | 85 | 77 | 70
  Week5 | -8.13 (2.02) | -13.97 (1.93) | -11.09 (2.01) | -6.62 (2.03)
  Week6: number analyzed (Participants) | 73 | 81 | 68 | 70
  Week6 | -8.26 (2.10) | -14.95 (2.00) | -11.49 (2.10) | -7.63 (2.11)

2. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Positive Subscale Score.
Description: PANSS consisted of three subscales: a total of 30 symptom constructs. For each construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness, and hostility. The PANSS positive subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Number analyzed (Participants) | 112 | 113 | 109 | 113
units on a scale
  Week1: number analyzed (Participants) | 110 | 112 | 109 | 113
  Week1 | -0.96 (0.36) | -1.31 (0.36) | -0.70 (0.36) | -1.09 (0.35)
  Week2: number analyzed (Participants) | 94 | 104 | 97 | 98
  Week2 | -1.72 (0.45) | -2.31 (0.44) | -1.61 (0.45) | -2.25 (0.44)
  Week3: number analyzed (Participants) | 86 | 97 | 88 | 85
  Week3 | -2.07 (0.52) | -3.21 (0.51) | -2.71 (0.52) | -2.57 (0.52)
  Week4: number analyzed (Participants) | 80 | 92 | 82 | 77
  Week4 | -2.39 (0.57) | -3.69 (0.54) | -3.09 (0.56) | -2.90 (0.56)
  Week5: number analyzed (Participants) | 76 | 85 | 77 | 70
  Week5 | -2.19 (0.62) | -4.05 (0.60) | -2.89 (0.62) | -3.26 (0.63)
  Week6: number analyzed (Participants) | 73 | 81 | 68 | 70
  Week6 | -2.22 (0.64) | -4.32 (0.61) | -3.15 (0.64) | -3.69 (0.64)

3. Secondary Outcome: Mean Change From Baseline to Week 6 in PANSS Negative Subscale Score.
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS negative subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: EEfficacy sample（FAS : Full Analysis Set） consisted of all participants who received at least one dose of study medication and have Baseline and at least one Post-Baseline PANSS total score evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Number analyzed (Participants) | 112 | 113 | 109 | 113
units on a scale
  Week1: number analyzed (Participants) | 110 | 112 | 109 | 113
  Week1 | -0.54 (0.27) | -0.83 (0.27) | -0.71 (0.27) | -0.59 (0.27)
  Week2: number analyzed (Participants) | 94 | 104 | 97 | 98
  Week2 | -1.08 (0.37) | -1.46 (0.36) | -1.76 (0.36) | -0.72 (0.36)
  Week3: number analyzed (Participants) | 86 | 97 | 88 | 85
  Week3 | -1.64 (0.41) | -2.41 (0.39) | -2.27 (0.40) | -1.14 (0.40)
  Week4: number analyzed (Participants) | 80 | 92 | 82 | 77
  Week4 | -2.36 (0.46) | -2.90 (0.44) | -2.94 (0.46) | -0.81 (0.46)
  Week5: number analyzed (Participants) | 76 | 85 | 77 | 70
  Week5 | -2.31 (0.52) | -3.24 (0.50) | -3.19 (0.52) | -0.85 (0.52)
  Week6: number analyzed (Participants) | 73 | 81 | 68 | 70
  Week6 | -2.34 (0.55) | -3.48 (0.52) | -3.24 (0.55) | -1.20 (0.55)

4. Secondary Outcome: Mean Change From Baseline to Week 6 in Clinical Global Impression-Severity of Illness (CGI-S)
Description: Severity of illness for each participant was rated using the CGI-S, which was the secondary efficacy endpoint. To perform this assessment, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Number analyzed (Participants) | 112 | 113 | 109 | 113
units on a scale
  Week1: number analyzed (Participants) | 111 | 112 | 109 | 113
  Week1 | -0.13 (0.06) | -0.18 (0.06) | -0.09 (0.06) | -0.15 (0.06)
  Week2: number analyzed (Participants) | 95 | 104 | 97 | 98
  Week2 | -0.26 (0.08) | -0.36 (0.08) | -0.34 (0.08) | -0.25 (0.08)
  Week3: number analyzed (Participants) | 86 | 97 | 88 | 85
  Week3 | -0.38 (0.09) | -0.52 (0.09) | -0.50 (0.09) | -0.36 (0.09)
  Week4: number analyzed (Participants) | 81 | 92 | 82 | 77
  Week4 | -0.48 (0.09) | -0.62 (0.09) | -0.50 (0.09) | -0.40 (0.09)
  Week5: number analyzed (Participants) | 76 | 85 | 77 | 70
  Week5 | -0.45 (0.11) | -0.81 (0.10) | -0.56 (0.10) | -0.52 (0.11)
  Week6: number analyzed (Participants) | 73 | 81 | 68 | 70
  Week6 | -0.52 (0.11) | -0.85 (0.11) | -0.62 (0.11) | -0.57 (0.11)

5. Secondary Outcome: Mean Clinical Global Impression-Improvement (CGI-I) Scale Score at Week 6.
Description: The efficacy of trial medication was rated for each participant using the CGI-I. The study physician would rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition at Baseline prior to the first dose of double-blind study medication. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Number analyzed (Participants) | 112 | 113 | 109 | 113
units on a scale
  Week1: number analyzed (Participants) | 111 | 112 | 109 | 113
  Week1 | 3.87 (0.92) | 3.84 (0.96) | 4.01 (0.93) | 3.92 (1.04)
  Week2 | 3.87 (1.10) | 3.68 (1.02) | 3.79 (1.13) | 3.88 (1.26)
  Week3 | 3.89 (1.20) | 3.53 (1.04) | 3.77 (1.20) | 3.92 (1.36)
  Week4 | 3.83 (1.23) | 3.51 (1.16) | 3.81 (1.23) | 3.90 (1.36)
  Week5 | 3.92 (1.27) | 3.42 (1.23) | 3.76 (1.30) | 3.86 (1.48)
  Week6 | 3.90 (1.32) | 3.49 (1.30) | 3.78 (1.33) | 3.83 (1.49)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 30 days after the last dose of study medication.
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/114 | 0/113 | 0/116
Serious Adverse Events (participants affected / at risk) | 8/115 | 5/114 | 5/113 | 5/116
Other Adverse Events (participants affected / at risk) | 49/115 | 46/114 | 49/113 | 56/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1mg (N=115) | Brexpiprazole 2mg (N=114) | Brexpiprazole 4mg (N=113) | Placebo (N=116)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Electroencephalogram abnormal (Investigations) | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 7 | 5 | 4 | 5
Psychiatric symptom (Psychiatric disorders) | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1mg (N=115) | Brexpiprazole 2mg (N=114) | Brexpiprazole 4mg (N=113) | Placebo (N=116)
Constipation (Gastrointestinal disorders) | 8 | 8 | 7 | 9
Vomiting (Gastrointestinal disorders) | 7 | 5 | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 6 | 2
Nausea (Gastrointestinal disorders) | 4 | 6 | 3 | 2
Dental caries (Gastrointestinal disorders) | 6 | 0 | 4 | 1
Nasopharyngitis (Infections and infestations) | 12 | 8 | 10 | 11
Blood prolactin increased (Investigations) | 1 | 3 | 7 | 3
Headache (Nervous system disorders) | 8 | 9 | 3 | 5
Akathisia (Nervous system disorders) | 2 | 4 | 6 | 8
Schizophrenia (Psychiatric disorders) | 20 | 13 | 23 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No